CLINICAL TRIAL: NCT07122869
Title: Eligibility of Patients Referred to Emergency Departments by Their General Practitioners for Care in Walk-in Clinics: A Single-Center Study in Île-de-France
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0115_URGENCES
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Emergency Service, Hospital; Primary Health Care; General Practitioners; Walk-In Clinics; Patient Admission; Health Services Accessibility
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to find out how many patients sent to the emergency department by their general practitioner could instead be treated in a walk-in clinic. Walk-in clinics provide quick, basic medical care without an appointment and can perform simple tests like blood work and X-rays. By identifying patients who don't need full hospital emergency care, this study hopes to improve patient flow and reduce overcrowding in emergency rooms in the Île-de-France region.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient referred to the emergency department (ED) with a letter from a general practitioner (GP)
* ED visit during the study hours (Monday to Friday, 9 a.m. to 8 p.m.)
* Consultation in the selected adult emergency service
* Medical or traumatic reason justifying the ED visit
* Patient stable at arrival and during ED care

Exclusion Criteria:

* Patients under 18 years old (pediatric cases excluded)
* No referral letter or proof of GP referral
* ED visit outside study hours (weekends, nights)
* Patients requiring intensive hospital care defined by:
* Intravenous treatments (e.g., antibiotics, fluids)
* Heavy imaging exams (CT scan, MRI) during the visit
* Diagnoses with immediate life- or function-threatening conditions (e.g., myocardial infarction, stroke, severe infection)
* Hospitalization decided during or after ED visit
* Clinical instability at or during ED visit (abnormal vital signs, respiratory distress, etc.)
* Patients referred for non-medical reasons (social issues, lack of medical follow-up)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from adult patients who visit the emergency department of a single hospital in Île-de-France between July 2023 and July 2025. Specifically, they must have been referred to the emergency department by their general practitioner with a referral letter and have visited during weekdays between 9 a.m. and 8 p.m. Only patients who are medically stable at arrival and have a medical or traumatic reason for their visit will be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Referred by General Practitioners to the Emergency Department Who Could Have Been Managed in a Walk-in Clinic | 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Gonesse, Gonesse, France, France